CLINICAL TRIAL: NCT05660863
Title: A Bridged Phase 1, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Multiple Dose of MN-08 in Healthy Subjects
Brief Title: A Multiple Dose Study to Investigate Safety, Tolerability and Pharmacokinetics of MN-08 Tablets
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Magpie Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21607
Record Dates: First submitted 2022-12-01; First posted 2022-12-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- cohort 1：MN-08 24 mg/day (Experimental): 2 x 6 mg MN-08 tablets for a total dose of 12 mg or 2 matching placebo tablets (given approximately every 12 hours) for 6.5 consecutive days, until the morning dose of Day 7.
  Interventions: Drug: MN-08 24 mg/day
- cohort 2：MN-08 60 mg/day (Experimental): 5 x 6 mg MN-08 tablets for a total dose of 30 mg or 5 matching placebo tablets (given approximately every 12 hours) for 6.5 consecutive days, until the morning dose of Day 7.
  Interventions: Drug: MN-08 60 mg/day

INTERVENTIONS:
Drug: MN-08 24 mg/day — Subjects in this cohort will receive 12 mg MN-08 tablets b.i.d. for a total daily dose of 24 mg or matching placebo for 6 consecutive days, and the last dose (12 mg) on the morning of Day 7.
  Arms: cohort 1：MN-08 24 mg/day
Drug: MN-08 60 mg/day — Subjects in this cohort will receive 30 mg MN-08 tablets b.i.d. for a total daily dose of 60 mg or matching placebo tablets for 6 consecutive days, and the last dose (30 mg) on the morning of Day 7.
  Arms: cohort 2：MN-08 60 mg/day

SUMMARY:
This trial is a single-center, Phase 1, placebo-controlled, double-blind, multiple-dose study in two ascending dose cohorts of healthy subjects. The primary objective of the trial is to assess the safety and tolerability of multiple doses of MN-08 tablet administered for 6.5 consecutive days in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be included in the study:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥ 18 and ≤ 45 years of age, with body mass index (BMI) > 18.0 and < 30.0 kg/m2 , and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to the first dosing. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Investigator.
   2. the absence of a clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Female subjects must not be pregnant, breastfeeding, or at risk to become pregnant during study participation. Female subjects must have a negative serum pregnancy test at screening (within 72 hours of the first dose of study medication) if of childbearing potential, or be of non-childbearing potential. Non-childbearing potential is defined as:

   1. post-menopausal female (absence of menses for 12 months prior to the first study drug administration, or having had a bilateral oophorectomy, or hysterectomy with bilateral oophorectomy at least 6 months prior to the first study drug administration); or
   2. surgically sterile female (hysterectomy or tubal ligation at least 6 months prior to drug administration).
4. Female subjects of childbearing potential (childbearing potential defined as not post menopausal nor surgically sterile) must agree to use a reliable method of birth control (see below for details) or remain abstinent during the study, starting with the screening visit until at least 90 days after the last study drug administration.
5. Male subjects who have not been vasectomized for at least 6 months, and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods from the first study drug administration until at least 90 days after the last study drug administration:

   1. simultaneous use of a male condom and, for the female partner, hormonal contraceptives used since at least 4 weeks prior or intra-uterine contraceptive device placed since at least 4 weeks prior to study.
   2. simultaneous use of a male condom and, for the female partner, a diaphragm or cervical cap with intravaginally applied spermicide.
6. Male subjects (including men who have had a vasectomy) with a pregnant partner must agree to use a condom from the first study drug administration until at least 90 days after the last study drug administration.
7. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration
8. Capable of signing the informed consent form.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Subjects with any following clinical illness at screening, including but not limited to respiratory, circulatory, digestive, hematological, endocrine, immunological, dermatological, and ENT abnormalities.
3. Subjects with digestive, liver, or kidney diseases which could affect the pharmacokinetics of drugs.
4. Positive urine drug screen, alcohol breath test, or urine cotinine test at screening.
5. History of allergic reactions to MN-08 or other related drugs, or to any excipient in the formulation.
6. Positive pregnancy test at screening.
7. Clinically significant ECG abnormalities or vital sign abnormalities, including: systolic BP lower than 90 or over 139 mmHg, diastolic BP lower than 60 or over 89 mmHg, or HR less than 55 or over 100 bpm; orthostatic BP: decrease in systolic blood pressure of 20 mmHg or higher, decrease in diastolic blood pressure of 10 mmHg or higher, or increase in heart rate of 30 bpm or higher within 2 to 3 minutes after passing from a supine to a standing position at screening.
8. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
9. History of significant drug abuse within 1 year prior to screening, or use of soft drugs (such as marijuana) within 3 months prior to the screening visit, or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
10. Subjects drinking excessive amounts of tea, coffee, or caffeinated beverages (more than 8 cups,1 cup = 250 mL) every day before the screening, or those who cannot agree to prohibit drinking tea, coffee, and/or products containing caffeine, grapefruit, or poppy 24 hours before dosing and during the study period.
11. Smoking history of 5 cigarettes per day within 3 months before the study, or those who cannot stop smoking 24 h before dosing and during the study period.
12. Have undergone major surgery 6 months before the study, or plan to have surgery during the study.
13. Have been vaccinated within 3 months prior to the study.
14. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
15. Use of medications for the time frames specified below, except for medications prescribed by the Investigator on a case-by-case basis because they have been judged unlikely to affect the pharmacokinetic profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. Prescription medications within 14 days prior to the first dosing.
    2. Over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing, except for the occasional use of acetaminophen (up to 2 g daily).
    3. Depot injection or implantation of any drug within 3 months prior to the first dosing.
    4. Any drugs known to induce or inhibit hepatic drug metabolism (including St. John's Wort) within 30 days prior to the first dosing.
16. Donation of plasma within 7 days prior to dosing. Donation or blood loss (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
17. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.
18. Breastfeeding subject.
19. Any history of suicidal ideation or suicidal behavior (within 2 years prior to screening), as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS; baseline version).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs and SAEs | Through study completion, an average of 12 days
  Incidence and severity of treatment emergent adverse events (TEAEs) and Serious Adverse Events (SAEs) after multiple doses of MN-08 administered for 6.5 consecutive days in healthy subjects.
Incidence and severity of treatment-related adverse events | Through study completion, an average of 12 days
  Incidence and severity of treatment-related adverse events determined by changes from screening (baseline) of findings from vital signs, ECG, and clinical laboratory parameters per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Single dose peak plasma concentration (Cmax) for MN-08 | Pre dose and up to 12 hours post dose after the morning dosing of Day 1.
  Peak plasma concentration (Cmax) for MN-08 after single oral doses of MN-08 tablets.
Single dose area under the plasma concentration versus time curve (AUC) for MN-08 | Pre dose and up to 12 hours post dose after the morning dosing of Day 1.
  Area under the plasma concentration versus time curve (AUC) for MN-08 after single oral doses of MN-08 tablets.
Single dose time to peak plasma concentration (Tmax) for MN-08 | Pre dose and up to 12 hours post dose after the morning dosing of Day 1.
  Time to peak plasma concentration (Tmax) for MN-08 after single oral doses of MN-08 tablets.
Repeated dose peak plasma concentration (Cmax) for MN-08 | Pre dose and up to 120 hours post dose after the morning dosing of Day 7.
  Peak plasma concentration (Cmax) for MN-08 after multiple oral doses of MN-08 tablets.
Repeated dose steady-state plasma concentration (Css) for MN-08 | Pre dose and up to 120 hours post dose after the morning dosing of Day 7.
  Steady-state concentration (Css) for MN-08 after multiple oral doses of MN-08 tablets.
Repeated dose area under the plasma concentration versus time curve (AUC) for MN-08 | Pre dose and up to 120 hours post dose after the morning dosing of Day 7.
  Area under the plasma concentration versus time curve (AUC) for MN-08 after multiple oral doses of MN-08 tablets.
Repeated dose time to peak plasma concentration (Tmax) for MN-08 | Pre dose and up to 120 hours post dose after the morning dosing of Day 7.
  Time to peak plasma concentration (Tmax) for MN-08 after multiple oral doses of MN-08 tablets.
Repeated dose terminal elimination half-life (t1/2) for MN-08 in plasma | Pre dose and up to 120 hours post dose after the morning dosing of Day 7.
  Terminal elimination half-life (t1/2) for MN-08 after multiple oral doses of MN-08 tablets.
Repeated dose ratio of accumulation (RA) for MN-08 | Pre dose and up to 120 hours post dose after the morning dosing of Day 7.
  Ratio of accumulation (RA) for MN-08 after multiple oral doses of MN-08 tablets.